CLINICAL TRIAL: NCT03736122
Title: A Phase I/IIa Study of Syngenon (BSG-001) for Inhalation in Subjects With Malignant Pleural Effusion and/or Malignant Ascites
Brief Title: A Study of Syngenon (BSG-001) for Inhalation in Subjects With Malignant Pleural Effusion and/or Malignant Ascites
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BioSyngen Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSG-001-001
Record Dates: First submitted 2018-10-30; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Malignant Pleural Effusion; Malignant Ascites
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BSG-001 (Experimental): Inhalation route, daily
  Interventions: Drug: BSG-001

INTERVENTIONS:
Drug: BSG-001 — BSG-001 is in solution form, 4mg per vial (2mg/mL) with Inhalation as route of administration using nebulizer.
  BSG-001 will be administrated as an approximately 5 - 30 minutes inhalation session daily for 3 cycles (in repeated 28 days cycle).

SUMMARY:
Malignant pleural effusion and/ or malignant ascites is generally defined by presence of malignant cells in the effusion fluid. The first-line therapies are mostly intrusive, medically demanding and inefficient, and therefore, it is important to study and develop new therapeutic option to address the unmet need.

This protocol for BSG-001 is developed for the treatment of malignant pleural effusion and/ or malignant ascites. BSG-001 is an immune-modulator primarily exerts its effect via Toll-like receptor.

The purpose of this study is to assess the safety and tolerability of BSG-001. All eligible subjects will receive BSG-001 for at least 12 weeks (3 cycles).

DETAILED DESCRIPTION:
This study is a phase 1/2a, single arm study with main purpose to evaluate the safety, tolerability and efficacy of BSG-001 in subjects with cancer that causes an abnormal amount of fluid to collect between the thin layers of tissue (pleura) lining the outside of the lung and the wall of the chest cavity, namely malignant pleural effusion and/ or subjects with cancer that causes the accumulation of fluid in the peritoneal cavity, causing abdominal swelling, namely malignant ascites.

The study aims to recruit 9 - 18 subjects in phase 1, and once the safety, tolerability and the preliminary efficacy of BSG-001 reach an optimal target exposure for recommended dose (RD), phase 2a will be opened for enrolment of approximately 40 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented malignant pleural effusion and/or malignant ascites OR morphological diagnosis of malignant pleural effusion and/or malignant ascites by CT or ultrasound
2. Histologically confirmed cancer
3. Malignant pleural effusion and/or malignant ascites clinically judged as not responsive to conventional systemic therapy(ies) for primary malignancy
4. Adequate liver and renal function as defined below:
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. Life expectancy of > 12 weeks
7. Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures
8. Females of childbearing potential must have a negative serum pregnancy test at screening and be willing to have additional serum pregnancy tests during the study.
9. Willing and able to comply with all study procedures

Exclusion Criteria:

1. Presence of > grade 3 active infection or gastric bleeding at the time of screening
2. Change in chemotherapy regimen within 28 days before Day 1 of study drug administration
3. Concurrent use of any investigational product (IP) or investigational medicine within 28 days before Day 1 of study drug administration
4. Symptomatic interstitial lung disease or inflammatory pneumonitis
5. Concurrent disease or condition which, in the opinion of the Investigator, would pose a risk to patient safety or interfere with study participation or interpretation of individual patient results
6. Breastfeeding at screening or planning to become pregnant (self or partner) at any time during study participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of BSG-001 assessed with incidence of Treatment-Emergent Adverse Events (AEs) and Serious AEs | From start of treatment throughout 12 weeks dosing
  Treatment-Emergent Adverse Events (AEs) and Serious AEs will be assessed by CTCAE v4.0 or higher version
Efficacy of BSG-001 assessed with change in fluid volume of Malignant Pleural Effusion and/or Malignant Ascites | From start of treatment throughout 12 weeks dosing, until disease progression and onward survival follow up up to 6 months or study completion, whichever came first.
  Efficacy of BSG-001 will be assessed with change in frequency and total change volume (for subjects require paracentesis and/or thoracentesis) and assessed by radiographic imaging (CT/ ultrasound) (for subjects without catheter drainage)

SECONDARY OUTCOMES:
Recommended dose (RD) of BSG-001 | Start of treatment throughout 28-day DLT dosing period
  RD will be assessed with incidence of BSG-001-related Adverse Events Grading during the dose limiting toxicity (DLT) period

OTHER OUTCOMES:
Subjects' reported quality of life [European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTCQLQ-30), version 3] | From screening/ baseline, followed by Day 1 of every cycle prior to other procedures (each cycle is 28 days) for 3 cycles.
  Reported quality of life will be assessed through EORTC QLQ-30 questionnaire score change from baseline, by a four-point scale (first 28 questions) and a 7-point scale (last 2 questions) total of 30 questions, where higher score represents higher (better) response level. Calculation is based on linear transformation to standardise the raw score, so that scores range from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Lietao Li, MD, Study Director — BioSyngen Australia Pty Ltd
Locations (1):
- Flinders Medical Centre, Adelaide, South Australia, Australia